CLINICAL TRIAL: NCT02940080
Title: Effect of Anthocyanins Extracted From Purple Potatoes on Healthy Study Subjects' Postprandial Glycemia and Insulinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Principal Investigator, University of Turku
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Siniset perunat 2
Record Dates: First submitted 2016-10-13; First posted 2016-10-20 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Postprandial Glycemia
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anthocyanins and yellow potato (Experimental): 168 mg of anthocyanins extracted from purple-fleshed potatoes added to 350 g of steam-cooked mashed potatoes in water
  Interventions: Other: Dietary
- Yellow potato (Experimental): 350 g of steam-cooked mashed potatoes in water
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary

SUMMARY:
A randomized, single-blind cross-over clinical nutrition trial will be conducted. The effects of yellow-fleshed potatoes and yellow-fleshed potatoes supplemented with anthocyanins extracted from purple-fleshed potatoes on healthy men's postprandial glycemia and insulinemia will be compared. Additionally, the postprandial metabolism and metabolites, and the appearance and metabolism of the flavonoids and their metabolites is studied in plasma, urine and feces.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Male
* No regular medication
* No participation in a drug trial or blood donation within 2 months
* Non-smoker
* Signs informed consent
* Body mass index 18.5-27 kg/m2
* Fasting plasma cholesterol < 5.5 mmol/l
* Fasting plasma triacylglycerols < 2.6 mmol/l
* Fasting plasma glucose 4-6 mmol/l
* blood pressure <140/80 mmHg
* hemoglobin>130 g/l
* Fasting plasma alanine amino transferase (ALAT) <60 U/l (normal liver function)
* Fasting plasma thyroid-stimulating hormone (TSH) 0.4 - 4.5 mU/l (normal thyroid function)
* Fasting plasma creatinine <118 µmol/l (normal kidney function)

Exclusion Criteria:

* Regular smoking
* Alcohol abuse
* Regular medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma glucose concentration | 0min, 20min, 40min, 60min, 90min, 120min, 180min, 240min
Plasma insulin concentration | 0min, 20min, 40min, 60min, 90min, 120min, 180min, 240min

SECONDARY OUTCOMES:
Concentrations and quality of metabolites and flavonoid color compounds and their metabolites in plasma (NMR and (U)HPLC-MS/MS measurements) | 0min, 20min, 40min, 60min, 90min, 120min, 180min, 240min
Concentrations and quality of metabolites and flavonoid color compounds and their metabolites in urine (NMR and (U)HPLC-MS/MS measurements) | Before meal, and 0-4h, 4-8h, 8-16h, 16-24 h
Concentrations and quality of metabolites and flavonoid color compounds and their metabolites in feces (NMR and (U)HPLC-MS/MS measurements) | before and after meal
Area under the glucose concentration curve (AUC) | 0min, 20min, 40min, 60min, 90min, 120min, 180min, 240min
Area under the insulin concentration curve (AUC) | 0min, 20min, 40min, 60min, 90min, 120min, 180min, 240min

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa M Linderborg, PhD, Principal Investigator — Department of Biochemistry, University of Turku
Locations (1):
- Department of Biochemistry, University of Turku, Turku, Finland